CLINICAL TRIAL: NCT06385444
Title: Effects of Implantation Failure and Pregnancy Loss After in Vitro Fertilization on Couples' Psychological Stress
Brief Title: IVF Failure and Pregnancy Loss on Couples' Psychological Stress
Status: Not yet recruiting | Type: Observational
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-HS-020
Record Dates: First submitted 2024-04-17; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Fertilization in Vitro; Pregnancy Loss; Psychological Stress; Post-traumatic Stress
Keywords: IVF failure; IVF pregnancy Loss; Psychological Stress; Post-traumatic Stress; Anxiety and depression
MeSH Terms: conditions — Stress, Psychological; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The female spouse of a couple: Women in couples with IVF pregnancy loss and IVF failure
- The male spouse of a couple: Men in couples with IVF pregnancy loss and IVF failure

SUMMARY:
The goal of this observational study is to learn about The purpose of this study was to compare the psychological differences between couples after IVF transplant failure and IVF pregnancy loss, including the differences in anxiety, depression, stress and post-traumatic stress between women and their spouses. The main question it aims to answer is:

What are the psychological effects of IVF implantation failure and IVF pregnancy loss on women and the psychological differences between couples? Participants already taking IVF as part of their regular medical care will answer online survey questions about their joint pain for 1 years.

DETAILED DESCRIPTION:
The goal of this observational study is to learn about The purpose of this study was to compare the psychological differences between couples after IVF transplant failure and IVF pregnancy loss, including the differences in anxiety, depression, and stress between women and their spouses. Some couples will experience symptoms of post-traumatic stress reaction (PTS), and there are also large differences. The differences between couples discussed in this study also pay attention to male spouses. Guidance and education for male spouses can reduce cognitive differences between couples and generate understanding and empathy, which is conducive to promoting the stability of family relations and intimate relationships.

1. Does the number of IVF implant failures have a differential effect on anxiety, depression and fertility stress in women and their partners?
2. Does pregnancy loss after IVF transplantation have a differential effect on anxiety, depression, fertility stress and post-traumatic stress responses in women and their partners?

ELIGIBILITY:
Inclusion Criteria:

1. Couples who have undergone IVF at our center and have completed at least 1 embryo transfer.
2. Female age 20-45 years, male age 22-45 years.

Exclusion Criteria:

1. Couples with contraindications to pregnancy.
2. Couples who undergo donor IVF.
3. Infertility women caused by organic lesions.
4. Couples with previous mental disorders.

Ages: 20 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: The study was a prospective cohort study. The participants were from couples who underwent in vitro fertilization at the Reproductive Center of the First Hospital of Jilin University.Further questionnaires were conducted for couples with IVF failure and pregnancy loss
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
As the number of failed IVF implants increases, does it increase the difference in anxiety and depression between couples? | 1 year
  The questionnaires used were the Hospital Anxiety and Depression Scale (HADS). HADS was used to assess anxiety and depression symptoms. Each domain has seven items with score ranges of 0 to 3, and total scores of 0 to 21, with higher score indicates greater psychological stress.
  Compare whether there is a growing difference between couples as the number of IVF failures increases.
As the number of failed IVF implants increases, does it increase the difference in fertility stress between couples? | 1 year
  The questionnaires used were the Fertility Problem Inventory (FPI). The FPI contains 46 items in 5 psychometric domains that measure social concern，sexual concern, relationship concern, the need for parenthood, and rejection of a childfree lifestyle. The instrument uses a 6-point Likert scale (1=strongly disagree;6=strongly agree). A high score in the FPI indicates a high level of perceived fertility-related stress.
  Compare whether there is a growing difference between couples as the number of IVF failures increases.
Does pregnancy loss after IVF transplantation have a differential effect on anxiety and depression between couples? | 1 year
  The questionnaires used were the HADS. HADS was used to assess anxiety and depression symptoms. Each domain has seven items with score ranges of 0 to 3, and total scores of 0 to 21, with higher score indicates greater psychological stress.
  Compare whether there is a growing difference between couples with the extension of time after pregnancy loss(1 month, 3 months, 6 months).
Does pregnancy loss after IVF transplantation have a differential effect on post-traumatic stress responses between couples? | 1 year
  The questionnaires used were the Posttraumatic Stress Disorder Checklist-Civilian Version (PCL-C).
  PCL-C contains 17 items, with an overall symptom severity score out of 85, including 3 dimensions of re-experience, avoidance and hypervigilance. Each item was scored on a scale of 1 to 5(1= no reaction,5= extremely severe reaction). Higher score indicates greater Posttraumatic Stress.
  Compare whether there is a growing difference between couples with the extension of time after pregnancy loss(1 month, 3 months, 6 months).

CONTACTS AND LOCATIONS:
Overall Officials: Qi Xi, doctorate, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- the first hospital of Jilin University, Changchun, Jilin, China

REFERENCES:
- [Result] Zegers-Hochschild F, Adamson GD, Dyer S, Racowsky C, de Mouzon J, Sokol R, Rienzi L, Sunde A, Schmidt L, Cooke ID, Simpson JL, van der Poel S. The International Glossary on Infertility and Fertility Care, 2017. Hum Reprod. 2017 Sep 1;32(9):1786-1801. doi: 10.1093/humrep/dex234. PMID 29117321
- [Result] Vander Borght M, Wyns C. Fertility and infertility: Definition and epidemiology. Clin Biochem. 2018 Dec;62:2-10. doi: 10.1016/j.clinbiochem.2018.03.012. Epub 2018 Mar 16. PMID 29555319
- [Result] Agarwal A, Mulgund A, Hamada A, Chyatte MR. A unique view on male infertility around the globe. Reprod Biol Endocrinol. 2015 Apr 26;13:37. doi: 10.1186/s12958-015-0032-1. PMID 25928197
- [Result] Chachamovich JR, Chachamovich E, Ezer H, Fleck MP, Knauth D, Passos EP. Investigating quality of life and health-related quality of life in infertility: a systematic review. J Psychosom Obstet Gynaecol. 2010 Jun;31(2):101-10. doi: 10.3109/0167482X.2010.481337. PMID 20443659
- [Result] Cates W, Farley TM, Rowe PJ. Worldwide patterns of infertility: is Africa different? Lancet. 1985 Sep 14;2(8455):596-8. doi: 10.1016/s0140-6736(85)90594-x. PMID 2863605
- [Result] Khademi A, Alleyassin A, Amini M, Ghaemi M. Evaluation of sexual dysfunction prevalence in infertile couples. J Sex Med. 2008 Jun;5(6):1402-10. doi: 10.1111/j.1743-6109.2007.00687.x. Epub 2007 Dec 14. PMID 18086173
- [Result] Wischmann T. Implications of psychosocial support in infertility--a critical appraisal. J Psychosom Obstet Gynaecol. 2008 Jun;29(2):83-90. doi: 10.1080/01674820701817870. PMID 18484439
- [Result] Murphy FA. The experience of early miscarriage from a male perspective. J Clin Nurs. 1998 Jul;7(4):325-32. doi: 10.1046/j.1365-2702.1998.00153.x. PMID 9830973
- [Result] Facchinetti F, Matteo ML, Artini GP, Volpe A, Genazzani AR. An increased vulnerability to stress is associated with a poor outcome of in vitro fertilization-embryo transfer treatment. Fertil Steril. 1997 Feb;67(2):309-14. doi: 10.1016/S0015-0282(97)81916-4. PMID 9022608
- [Result] Cimadomo D, Craciunas L, Vermeulen N, Vomstein K, Toth B. Definition, diagnostic and therapeutic options in recurrent implantation failure: an international survey of clinicians and embryologists. Hum Reprod. 2021 Jan 25;36(2):305-317. doi: 10.1093/humrep/deaa317. PMID 33313697
- [Result] ESHRE Working Group on Recurrent Implantation Failure; Cimadomo D, de Los Santos MJ, Griesinger G, Lainas G, Le Clef N, McLernon DJ, Montjean D, Toth B, Vermeulen N, Macklon N. ESHRE good practice recommendations on recurrent implantation failure. Hum Reprod Open. 2023 Jun 15;2023(3):hoad023. doi: 10.1093/hropen/hoad023. eCollection 2023. PMID 37332387
- [Result] ESHRE Guideline Group on RPL; Bender Atik R, Christiansen OB, Elson J, Kolte AM, Lewis S, Middeldorp S, Mcheik S, Peramo B, Quenby S, Nielsen HS, van der Hoorn ML, Vermeulen N, Goddijn M. ESHRE guideline: recurrent pregnancy loss: an update in 2022. Hum Reprod Open. 2023 Mar 2;2023(1):hoad002. doi: 10.1093/hropen/hoad002. eCollection 2023. PMID 36873081
- [Result] Cumming GP, Klein S, Bolsover D, Lee AJ, Alexander DA, Maclean M, Jurgens JD. The emotional burden of miscarriage for women and their partners: trajectories of anxiety and depression over 13 months. BJOG. 2007 Sep;114(9):1138-45. doi: 10.1111/j.1471-0528.2007.01452.x. Epub 2007 Jul 26. PMID 17655731
- [Result] Farren J, Jalmbrant M, Falconieri N, Mitchell-Jones N, Bobdiwala S, Al-Memar M, Tapp S, Van Calster B, Wynants L, Timmerman D, Bourne T. Differences in post-traumatic stress, anxiety and depression following miscarriage or ectopic pregnancy between women and their partners: multicenter prospective cohort study. Ultrasound Obstet Gynecol. 2021 Jan;57(1):141-148. doi: 10.1002/uog.23147. PMID 33032364